CLINICAL TRIAL: NCT00564057
Title: Effects of Antihypertensive Treatment on Cardiac Remodelling and Metabolic Profile in HIV Infected Patients: Randomized Longitudinal Study With Candesartan Versus Lercanidipine
Brief Title: Effects of Antihypertensive Treatment in HIV Infected Patients: Candesartan Versus Lercanidipine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 44758
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-11

CONDITIONS: HIV Infections; Hypertension
Keywords: HIV; blood pressure; left ventricle; metabolic profile; treatment experienced
MeSH Terms: conditions — HIV Infections; Hypertension | interventions — candesartan; lercanidipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): candesartan 8-16 mg once daily
  Interventions: Drug: candesartan
- 2 (Active Comparator): lercanidipine 10-20 mg once daily
  Interventions: Drug: lercanidipine

INTERVENTIONS:
Drug: candesartan — tablet 8-16 mg once daily, one year
  Arms: 1
Drug: lercanidipine — tablets 10-20 mg once daily, one year
  Arms: 2

SUMMARY:
Human immunodeficiency virus infection and highly active antiretroviral therapy (HAART) are associated with an increased risk of cardiovascular disease: a wide range of alterations in lipid and glucose metabolism has been increasingly recognized in HIV patients treated with HAART. Few data are available on the effects of antihypertensive treatment on cardiac morpho-functional characteristics and metabolic parameters in HIV patients. Aim of the study is to assess the effects of chronic therapy with angiotensin receptor blocker(candesartan)or calcium channel blocker (lercanidipine)on metabolic profile and cardiac remodelling in HIV hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* office blood pressure > 140/90 mmHg
* no antihypertensive treatment
* good quality echocardiogram

Exclusion Criteria:

* cardiovascular diseases
* hypothyroidism
* diabetes
* secondary hypertension
* hepatic and renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-09; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
morpho-functional left ventricle characteristics | one year
metabolic profile | one year

SECONDARY OUTCOMES:
systolic and diastolic blood pressure | one year

CONTACTS AND LOCATIONS:
Overall Officials: anna maria grandi, MD, Study Chair — University of Insubria, Varese, ITALY; paolo grossi, MD, Principal Investigator — University of Insubria, Varese, Italy; andrea maria maresca, MD, Principal Investigator — University of Insubria, Varese, Italy; eleonora nicolini, MD, Principal Investigator — University of Insubria, Varese, Italy; massimo giola, MD, Principal Investigator — University of Insubria, Varese, Italy
Locations (1):
- University of Insubria, Department of Clinical Medicine, Varese, Italy

REFERENCES:
- [Background] Grinspoon SK. Metabolic syndrome and cardiovascular disease in patients with human immunodeficiency virus. Am J Med. 2005 Apr;118 Suppl 2:23S-28S. doi: 10.1016/j.amjmed.2005.01.047. PMID 15903292
- [Background] Gazzaruso C, Bruno R, Garzaniti A, Giordanetti S, Fratino P, Sacchi P, Filice G. Hypertension among HIV patients: prevalence and relationships to insulin resistance and metabolic syndrome. J Hypertens. 2003 Jul;21(7):1377-82. doi: 10.1097/01.hjh.0000059071.43904.dc. PMID 12817187
- [Background] Friis-Moller N, Sabin CA, Weber R, d'Arminio Monforte A, El-Sadr WM, Reiss P, Thiebaut R, Morfeldt L, De Wit S, Pradier C, Calvo G, Law MG, Kirk O, Phillips AN, Lundgren JD; Data Collection on Adverse Events of Anti-HIV Drugs (DAD) Study Group. Combination antiretroviral therapy and the risk of myocardial infarction. N Engl J Med. 2003 Nov 20;349(21):1993-2003. doi: 10.1056/NEJMoa030218. PMID 14627784
- [Background] Meng Q, Lima JA, Lai H, Vlahov D, Celentano DD, Strathdee S, Nelson KE, Tong W, Lai S. Use of HIV protease inhibitors is associated with left ventricular morphologic changes and diastolic dysfunction. J Acquir Immune Defic Syndr. 2002 Jul 1;30(3):306-10. doi: 10.1097/00126334-200207010-00006. PMID 12131567
- [Background] Lindholm LH, Persson M, Alaupovic P, Carlberg B, Svensson A, Samuelsson O. Metabolic outcome during 1 year in newly detected hypertensives: results of the Antihypertensive Treatment and Lipid Profile in a North of Sweden Efficacy Evaluation (ALPINE study). J Hypertens. 2003 Aug;21(8):1563-74. doi: 10.1097/01.hjh.0000084723.53355.76. PMID 12872052